CLINICAL TRIAL: NCT05473702
Title: Smart Textile Sensor System for Health Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanowear Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-90-0093
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Heart Disease Chronic; Pulmonary Disease, Chronic Obstructive; Blood Pressure; Heart Rhythm Disorder
Keywords: Remote health monitoring; Wearable monitoring; Respiration rate; Heart rate; Heart Sound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cardiac health subjects: Subjects over 18 years of age. Subject should satisfy any one of the following:
  * Healthy subject with no pre-existing conditions.
  * Subject with prehypertension
  * Subject with hypertension
  * Subject undergoing dialysis
  Interventions: Device: Nanowear SimpleSense Wearable monitoring device

INTERVENTIONS:
Device: Nanowear SimpleSense Wearable monitoring device — The Nanowear SimpleSense is a non-invasive, wearable and portable medical device for evaluation and monitoring of cardiopulmonary condition. It utilizes physiologic and biometric sensors, SAU, and software system with a suite of algorithms to monitor patient. The parameters include: two vectors of ECG, two vectors of impedance cardiography, thoracic impedance, respiration, heart sounds, and actigraphy and postures. The device is comprised of a wearable device made of an elastomeric harness comprising of active and passive Nanosensors, heart sound sensor, connector to electrically connect the sensors to SAU, it comprises of Inertial Measurement Unit, analog front end, processing unit, storage unit, power supply, and a wireless module, and a software system equipped with the suite of algorithms to monitor heart. The signals are recorded by SAU, transferred to the iPhone over Bluetooth, which later transfers the data to a secure website over an internet connection Wi-fi or mobile network.

SUMMARY:
The present study will investigate a set of biomedical sensors with a wireless data communication system and evaluate the sensors' recording quality. The sensors and wearable wireless system have been approved by Food and Drug Administration (FDA) for recording Electrocardiography (ECG), Trans Thoracic Impedance (TTI), Heart Sounds and Acitigraphy. The sensors and wireless system will be used along with conventional sensor systems (as intended to be used).

DETAILED DESCRIPTION:
Procedures involving people:

The sensors- electrodes, conductor channels and semi-conductor channels- are in direct contact (with the body) or indirect contact through a transient layer of polyimide or silicon rubber. The amplifiers will boost the microvolt signals into the range where they can be accurately digitized using analog to digital converter. Subsequently, a wireless data communication system will transmit and receive the digitized data and a personal computer (or other relevant device) will store and display the recorded data. The sensors used for measurement for bioimpedance will pass a modulated current of 1-5 mA (rms) at 30kHz to 100kHz through the skin into subject body. This system will be powered by a 3.7 V battery source. The sensor system(s) will draw power through this system. The sensor systems that will be used for this study are:

1. Reusable flat gold and nanowire (gold or platinum or titanium) electrodes for ECG, ICG, TTI, EEG, EOG, EMG measurement..
2. Reusable Nanotextured textile coated with a thin film of metal (gold or silver or platinum or titanium) electrodes for ECG, ICG, TTI, EEG, EOG, EMG measurement.
3. Reusable Heart sound sensor, amplifier circuitry, for heart sound measurement.
4. Reusable sensor, temperature dependent resistor circuitry, for body temperature measurement.
5. Reusable sensor, strain dependent resistor circuitry, for measurement of respiration effort.
6. Reusable sensor, piezoelectric circuitry, for blood pressure measurement.
7. Reusable acceleration and rotation detection sensor with respect to x,y,z axis. sensor, amplifier circuitry, for measurement of activity (actigraphy) of the subjects.
8. Reusable optoelectronic sensor, amplifier circuitry, for blood oxygen level measurement.
9. Reusable sensor, piezoelectric and optoelectronic circuitry, for pulse rate measurement.
10. A wearable wireless system: compact embedded systems and a portable battery, enclosed in a sturdy ebonite box.

The sensors will be fabricated on polyimide (KAPTON®) and polyester films, and textile fabric and will require to be mounted on subject's skin. This will be accomplished by using standard surgical waterproof tape or braces made form materials like polyester, nylon, silicone rubber sheetand textile fabric. At all times this polyimide or polyester material will be the only component in contact with test subject's skin. The sensor recordings will be taken from the test subjects in different physical states: supine position, sitting and relaxed, standing up and/or walking briskly, engaging in moderately rigorous exercise (not cardiovascular exercise).

1 Device specific protocols: 1.1 ECG measurements with Dry Electrodes:

1. Sit comfortably on a bed or chair
2. Mark the electrode position on the skin.
3. After cleaning skin, place electrodes into position with a brace.
4. Depending on the experiment design, the test subject may assume the said physical states (supine, sitting, standing, walking, moderate exercise).
5. Typical duration of test will last for 30 min- 1 hr.
6. The electrode positions, on the test subject, for real time ECG measurement will be as shown in figure 1. Electrodes 7, 8, 9 and 10 constitute the driven right leg Einthoven augmented lead system. Electrodes 1 through 6 are chest leads used as part of the standard 12 electrode system.

Figure 1: Electrode placement map for real time ECG signal acquisition. 1.2 Skin contact impedance measurement with Dry Electrodes:

The procedure will be carried out by a trained operator. The steps are as follows:

1. The subject will be asked to sit comfortably on a bed or chair.
2. The electrode positions will be marked on the arm.
3. After cleaning the skin, place the electrodes in position with the help of braces.
4. The electrodes are connected to the electrode impedance meter.
5. The impedance readings will be tabulated (manually) at intervals of up to 15 minute. The duration of the experiment will range from 60 to 90 minutes.

At regular intervals, the operator will ask the subject for any tingly feeling on subject's arm. This will serve as a precaution. However, the impedance meter (in use) is a dedicated device for measuring skin-electrode contact impedance.

1.3 Respiration Sensor: The respiration sensor has been fabricated with the device electronics on flexible substrates (films): polyimide (KAPTON ®), silicone rubber, poly ethylene napthalate. These sensors will be mounted on either elastic polyester strap or inelastic nylon strap. The only materials in direct contact with the skin will be the nylon/polyester band and silicone or KAPTON. The strap will have to be worn around the midriff where the effective increase and decrease in diameter is maximal during inhalation and exhalation respectively. All wires leading to the sensor will be commercially available insulated copper/nickel cables.

1.3.1 Procedure involving test subject:

1. The elastic/nylon strap will be worn by the subject around the lower abdomen as indicated in figure 2.

   Figure 2: Strategy for mounting the respiration sensor for real time respiration effort signal acquisition
2. The subject will be requested to perform the following patterns of breathing:

1. Short shallow breathes. 2. Deep breathes. 3. Hold breath after deep inhalation. 4. Hold breath after deep exhalation. 5. Normal breathes after different intervals ranging from 1 second to 10 seconds.

The above tests involving different patterns of breathing are intended to be an exhaustive in terms of all practically observed patterns of breathing. Also, these conditions comprehensively cover the physical states (supine, sitting, standing, walking, moderate exercise) described in the initial part of section 2. The signal acquisition time period will be subjective to the calibration experiment or the hypothesis being tested.

For the standardization of this sensor, commercially available respiration sensor will also be mounted simultaneously and measurements will be compared.

1.4 Body Temperature Sensor: This sensor will be used to measure the body temperature at the skin. Similar to the respiration sensor, the device circuitry will be on flexible substrate. The only material in contact with the skin of the test subject will be KAPTON®. The sensor will be packaged to electrically insulate it from subject's body. All wires leading to the sensor will be commercially available insulated copper/nickel cables.

1.4.1 Procedure involving test subject:

1. The sensor will be placed on the side of the test subject below the underarm (for Axial Temperature), on the chest above the sternum, back or face as shown in figure 3.
2. The subject will, also, be asked to wear a commercially available dry bulb temperature sensor on the skin in the regions highlighted in figure 3.

   Figure 3: Strategy for mounting the temperature sensor for real time signal acquisition.
3. The readings will be taken in indoor and outdoor settings.
4. Data acquisition will be done while the subject is in the physical states (supine, sitting, standing, walking, moderate exercise) mentioned in section 2.

1.5 Blood Pressure and Pulse Rate Sensor: This sensor will be used for measurement of arterial blood pressure and pulse rate, heart sound and blood oxygen level in a non-invasive fashion. The device circuitry comprises of MEMS microphone, piezoelectric or optoelectronic transducer(s) mounted on a polyimide (KAPTON ®) or polyester film. Optoelectronic components have energy dissipation of less than 0.5 Watt. MEMS microphone is an off the shelf electronic component operating on 1.8 to 3.3 V and drawing 180 to 250 µA. This film will be in contact with test subject's skin. The sensor will be mounted on subject's left forearm, sternum or back, as shown in figure 4. The sensor will be electrically insulated from subject's body. All wires leading to the sensor will be commercially available insulated copper/nickel cables.

1.5.1 Procedure involving test subject:

1. Prior to commencing the test, standard pulse rate and blood pressure and blood oxygen level readings will be taken with the help of commercial pulse oxymeter and blood pressure cuff.
2. The blood pressure, heart sound and pulse rate sensors will be mounted on left forearm, sternum or back of the subject (Figure 4).

   Figure 4: Strategy for mounting blood pressure and pulse rate sensor system
3. Pulse, blood oxygen level, heart sound and blood pressure data will be recorded while the subject is in the physical states (supine, sitting, standing, walking, moderate exercise).
4. During the test, the subject will be asked to wear the commercial Pulse oxymeter for real time comparison pulse rate and blood oxygen level values.

1.6 Bioimpedance measurement with Dry Electrodes

1. Sit comfortably on bed or chair
2. Mark electrode position on the skin
3. Place electrodes into position on the skin with a brace
4. Depending on the experiment design, the test subject may assume the said physical states (supine, sitting, standing, walking, moderate exercise).
5. Typical duration of the test will last for 15 minutes to 12 hours
6. The electrode positions, on the test subject , for real time bioimpedance measurement will be as shown in figure 5.
7. Bioimpedance measurement will be done by using 4 electrodes placed on the skin as shown in figure 5. A modulated current of 1-5 mA (rms) at 30kHz to 100kHz is passed through subject's body between two electrodes 1,4 or 5,8 and resulting change in biopotential is measured between two electrodes 2,3 or 4,6. Bioimpedance is measured by a conversion circuit which is part of the wireless data communication system. A similar 4 electrode placement will be done on the arm, forehead, neck, torso or leg region of subjects body based on the objective of study.

1.7 Heart Sound measurement with Heart sound sensor

1. Sit comfortably on bed or chair
2. Mark electrode position on the skin
3. Place Heart sound sensor into position on the skin with a brace
4. Depending on the experiment design, the test subject may assume the said physical states (supine, sitting, standing, walking, moderate exercise).
5. Typical duration of the test will last for 15 minutes to 12 hours
6. The sensor position 9, on the test subject , for real time bioimpedance measurement will be as shown in figure 5.

Figure 5 1.8 EEG, EOG and EMG measurement with Dry Electrodes

1. Sit comfortably on bed or chair
2. Mark electrode position on the skin
3. Place electrodes into position on the skin with a brace or with adhesive patches
4. During the test the subject will be asked to perform eye movements, jaw movements and relax with eyes closed for purpose of calibration of sensor system.
5. Depending on the experiment design, the test subject may assume the said physical states (supine awake, supine sleep, right and left lateral awake, right and left lateral sleep, sitting, standing, walking).
6. Typical duration of the test will last for 15 minutes to 12 hours
7. The electrode positions, on the test subject , for real time EEG, EOG, EMG measurement will be as shown in figure 6. Where EEG electrodes are place on the forehead region (band), EOG electrodes are placed around the eye(s) with a reference electrode on the mastoid bone on either side and EMG electrode pair ( 2 electrodes placed at least 2mm apart) on the chin.

Figure 6 1.9 Acceleration and rotation detection sensor for measurement of activity (actigraphy) of the subjects

1. Sit comfortably on bed or chair
2. Place acceleration and rotation detection sensor into position on the skin with a brace
3. Depending on the experiment design, the test subject may assume the said physical states (supine, sitting, standing, walking, moderate exercise).
4. Typical duration of the test will last for 15 minutes to 12 hours
5. The sensor position, on the test subject , for real time activity measurement will be as shown in figure 7.

Figure 7

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject with no pre-existing conditions.
* Subject with prehypertension
* Subject with hypertension
* Subject undergoing dialysis

Exclusion Criteria:

* Pregnant women
* Subjects with implantable cardiac devices (for example, pacemaker or internal cardioverter defibrillator).
* Subjects with arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 willing subjects evenly spread across age range, gender, BMI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10-23 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy against gold standard devices | 1 year
  Efficacy of SimpleSense Electrocardiograph (ECG) signals against a Holter monitor: Simultaneous ECG signal capture from SimpleSense and Holter monitor. Obtain correlation (with 95% confidence interval) between amplitudes of simultaneously recorded ECG signals from SimpleSense and ECG signals from Holter monitor.
Efficacy against gold standard devices | 1 year
  Efficacy of SimpleSense Impedance cardiograph (ICG) signals against gold standard: Simultaneous bioimpedance and ICG signal capture from SimpleSense and Bioimpedance recorder. Obtain correlation (with 95% confidence interval) between amplitudes of simultaneously recorded bioimpedance and ICG signals from SimpleSense and signals from Bioimpedance recorder.
Efficacy against gold standard devices | 1 year
  Efficacy of SimpleSense Heart Sound signals against gold standard devices: Simultaneous Heart Sound signal capture from SimpleSense and Digital Stethoscope. Obtain correlation (with 95% confidence interval) between amplitudes of simultaneously recorded Heart Sound signal capture from SimpleSense and Digital Stethoscope.
Efficacy against gold standard devices | 1 year
  Efficacy of SimpleSense Posture against gold standard devices: Simultaneous 3 axis accelerometer signal capture from SimpleSense and Visual record of posture change. Obtain correlation (with 95% confidence interval) between amplitudes of simultaneously recorded 3 axis accelerometer signal capture from SimpleSense and Visual record of posture change.

SECONDARY OUTCOMES:
Blood pressure algorithm build | 1 year
  Trained and validated algorithm (SimpleSense-BP Software Application) that can compute blood pressure through the metrics measured by the SimpleSense device: Simultaneous recording of signals from SimpleSense and BP measurement from Sphygmomanometer cuff. Training a multi-variate algorithm and testing it for accuracy on separate subject cohorts. The mean absolute difference (MAD) and mean absolute percentage difference (MAPD) calculated between measured blood pressure from the cuff and the estimated blood pressure form the algorithm.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clincept, Atlanta, Georgia
  - Maimonides Medical Center, Brooklyn, New York
  - Nanowear R&D, State College, Pennsylvania